CLINICAL TRIAL: NCT04223414
Title: Ability of Changes in Analgesia Nociception Index to Assess the Stroke Volume Effects of a Volume Expansion of 250ml of Crystalloid in the Operating Room. REVANI Trial
Brief Title: Ability of Changes in Analgesia Nociception Index to Assess the Stroke Volume Effects of a Volume Expansion of 250ml of Crystalloid in the Operating Room
Acronym: REVANI
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2019/23
Record Dates: First submitted 2020-01-06; First posted 2020-01-10 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Volume Expansion; Fluid Responsiveness
Keywords: volume expansion; fluid responsiveness; stroke volume; perioperative optimization; analgesia nociception index

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Analgesia Nociception Index (ANI) — ANI will be used to analyse the autonomic nervous system's response to volume expansion.
  ANI will be assessed during surgery, before during and after the volume expansion

SUMMARY:
Volume expansion is the cornerstone of perioperative hemodynamic optimization. The main objective of volume expansion is to increase and maximize stroke volume. Hemodynamic changes have an impact on the autonomic nervous system. The analysis of heart rate variability allows an exploration of the autonomic nervous system and could therefore provide information on the effect of volume expansion. The Analgesia Nociception Index (ANI) is an analgesia monitor based on the concept of heart rate variability. By deviating from its original use, the investigators wish to evaluate the ability of ANI to identify a response to volume expansion.

DETAILED DESCRIPTION:
Perioperative optimization is based on volume maximization using volume expansion. The main objective of volume expansion is to increase stroke volume. The Franck-Starling curve is schematically divided into two portions: a vertical portion which mean that an increase in preload secondary to volume expansion will induce an increase in stroke volume; and a flat portion where volume expansion will not induce an increase in stroke volume. Perioperative optimization is based on stroke volume maximization using volume expansion.

In case of hypovolemia, there is a compensatory sympathetic stimulation with parasympathetic withdrawal. Volume expansion will lead to an increase in venous return and therefore in cardiac output, which will result in a decrease in sympathetic tone. The autonomic nervous system is therefore directly affected by these load changes. The analysis of heart rate variability, which has been studied for several years in various setting, allows the assessment of autonomic nervous system, through monitoring of the electrocardiogram. Experimental and clinical studies report the ability of variations in heart rate variability to detect a situation of hypovolemia. In anaesthesia, heart rate variability is used to evaluate the nociception-antinociception balance. Indeed, any nociceptive stimulation leads to an increase in sympathetic tone. MetroDoloris has developed a non-invasive monitor that provides an index, the Analgesia Nociception Index (ANI), to evaluate the nociception-antinociception balance by analysing the autonomic nervous system.

In this study, the original use of ANI will be diverted from its initial use, to analyse the autonomic nervous system's response to volume expansion. Thus, the aim of the present study is to determine whether a change in Analgesia Nociception Index can track the stroke volume effects of a volume expansion using 250ml of crystalloid in the operating room.

The follow up will be restricted to the duration of surgical intervention. The last data will be collected 5 minutes after the end of volume expansion.

ELIGIBILITY:
Inclusion Criteria:

* patient older than 18 years
* patient scheduled for neurosurgery in prone position
* patient equipped from an arterial catheter and stroke volume monitoring
* Patient for whom volume expansion is needed.

Exclusion Criteria:

* emergency surgery,
* cardiac dysfunction,
* arrythmia,
* beta-blockade therapy,
* pacemaker,
* intracranial hypertension,
* pregnancy,
* dysautonomia

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient scheduled for neurosurgery
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2020-01-29 (Actual); Primary Completion 2020-06-25 (Actual); Study Completion 2020-06-25 (Actual)

PRIMARY OUTCOMES:
ANI value variation (%) before and after the volume expansion | 5 minutes after volume expansion
  Changes in the analgesia nociception index during a volume expansion of 250 mL crystalloid during 10 minutes in patients who responded to volume expansion (stroke volume increase by 10% or more after volume expansion) and in patients who did not respond to volume expansion (stroke volume increase less than 10% after volume expansion).

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] de Courson H, Chadefaux G, Abel B, Georges D, Verchere E, Biais M. Ability of the Analgesia Nociception Index variations to identify a response to a volume expansion of 250 mL of crystalloids in the operating room (REVANI): a prospective observational study. BMC Anesthesiol. 2023 Jun 21;23(1):218. doi: 10.1186/s12871-023-02181-2. PMID 37344801